CLINICAL TRIAL: NCT03868150
Title: Assessment of Intra-Operative Atrial Fibrillation Inducibility As a Screening Tool to Prevent Post-Operative Atrial Fibrillation With Prophylaxis Amiodarone
Brief Title: Prevention of Postop Atrial Fibrillation Through Intraoperative Inducibility of Atrial Fibrillation and Amiodarone Treatment
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anson M Lee, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 38527
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Atrial Fibrillation
MeSH Terms: interventions — Amiodarone

STUDY DESIGN:
Intervention Model Description: Prospective randomized control trial of Amiodarone versus standard of care in patients with intraoperative inducible atrial fibrillation undergoing non emergent first-time cardiac surgery.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Inducible Atrial Fibrillation (Active Comparator): Treatment with Amiodarone
  Interventions: Drug: Amiodarone Injection; Device: Intraoperative Rapid Atrial Pacing
- Inducible Atrial Fibrillation - Standard Care (Other): No initial Amiodarone Treatment unless POAF seen on post operative care unit.
  Interventions: Drug: Amiodarone Injection; Device: Intraoperative Rapid Atrial Pacing
- Non-Inducible Atrial Fibrillation (Other): Amiodarone treatment if POAF seen on post-operative care unit
  Interventions: Device: Intraoperative Rapid Atrial Pacing

INTERVENTIONS:
Drug: Amiodarone Injection — Patients stratified into the amiodarone study group were administered amiodarone until day of discharge. Amiodarone administration began intraoperatively with the administration of a 150 mg IV amiodarone loading bolus prior to separation from coronary pulmonary bypass, followed by 1 mg/min IV amiodarone for six hours (360 mg), then 0.5 mg/min IV amiodarone for 18 hours (540 mg), then transitioned to 400 mg oral amiodarone twice a day until discharge. In total, patients in the amiodarone treatment group received 1,050mg of IV amiodarone plus 800mg/day of oral amiodarone thereafter until discharge.
  Arms: Inducible Atrial Fibrillation; Inducible Atrial Fibrillation - Standard Care
Device: Intraoperative Rapid Atrial Pacing — Intraoperative rapid atrial pacing for 30 seconds after cannulation and prior to initiation of cardiopulmonary bypass by having the surgeon attach insulated forceps to the superior right atrial free wall and connected to a temporary pacemaker to burst pace at a rate of 800 bpm for 30 seconds (pulse width 1.0 ms, output: 20 mA) Patients are monitored for successful atrial fibrillation induction defined as 30 seconds of sustained atrial fibrillation on ECG.

SUMMARY:
Patients undergoing first time cardiac surgery will undergo rapid atrial pacing prior to initiation of cardiopulmonary bypass to screen for AF inducibility. Patients with inducible AF will be randomized to prophylactic amiodarone treatment versus no treatment. Patients who are not inducible to AF will be treated with standard post-operative care. Patients will be monitored post-operatively to explore the value of intraoperative inducibility of AF to predict POAF and to evaluate whether the combination of intraoperative inducibility and precision amiodarone therapy is effective at reducing the incidence of POAF

DETAILED DESCRIPTION:
In the operating room, as part of the open heart surgery, the surgeon will stimulate the superior right atrium section of the heart with a pacemaker for 30 seconds just prior to starting the heart and lung bypass machine. The stimulation is done to see how sensitive the heart is to developing atrial fibrillation. This test result will be documented. The procedure will only take 60 seconds out of the entire operation. It does not involve taking any samples of tissue or blood. Following this step, if the heart demonstrates atrial fibrillation for at least 30 seconds then the participant will then be randomized to either receive the prophylactic drug treatment using Amiodarone or to no prophylactic drug administration. The participant has a 50% chance of receiving the FDA approved study drug Amiodarone. The study arms consist of prophylactic drug administration with Amiodarone, No prophylactic drug administration, or no atrial fibrillation reaction after stimulation with the pacemaker. The remainder of the surgical procedure will not be affected, and will follow routine surgical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for first-time non-emergent open-heart surgery for coronary artery bypass graft (CABG) revascularization, valvular repair or replacement, combined CABG with valve repair or replacement, or valve sparing aortic root repair
* Normal sinus rhythm
* No documented history of atrial fibrillation

Exclusion Criteria:

* Prior surgical procedures involving heart surgery and cardiopulmonary bypass
* Any prior documented history of atrial fibrillation, atrial flutter or atrial tachycardia lasting longer than 30 seconds
* Prior history of Amiodarone treatment for the management of supraventricular tachy-arrhythmias
* Patients requiring surgical treatment of atrial arrhythmias such as pulmonary vein isolation or Maze procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Decreasing the incidence of Post-Operative Atrial Fibrillation for Cardiac Surgery Patients | 30 days
  Identify predictors of developing atrial fibrillation in the hope of decreasing post-operative length of stay, the need for anticoagulation, decrease risk of stroke, DVT, and bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Anson Lee, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Derived] Pong T, Cyr K, Niesen J, Aparicio-Valenzuela J, Carlton C, Fischbein MP, Woo YJ, Boyd JH, Lee AM. Screening and Prophylactic Amiodarone Reduces Post-Operative Atrial Fibrillation in At-Risk Patients. J Am Coll Cardiol. 2020 Mar 24;75(11):1361-1363. doi: 10.1016/j.jacc.2020.01.016. No abstract available. PMID 32192666